CLINICAL TRIAL: NCT06321419
Title: Effects of Advanced Trauma Life Support® Training Compared to Standard Care on Adult Trauma Patient Outcomes: A Cluster Randomised Trial
Brief Title: Effects of Advanced Trauma Life Support® on Adult Trauma Patient Outcomes
Acronym: ADVANCE TRAUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The George Institute (Other)
Responsible Party: Principal Investigator, Martin Gerdin, Principal Researcher, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: atls-vs-standard-care
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Wounds and Injuries
Keywords: Advanced Trauma Life Support; Mortality; Disability; Return to work; Quality of Life
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Batched stepped-wedge cluster randomised trial. We will roll out the interventions to 30 clusters over six batches, so there will be five clusters in each batch. The clusters in each batch will be randomised to one of five implementation sequences, with one hospital randomised to each implementation sequence. All clusters will transition through three phases, first a standard care phase, then a one month transition phase during which the training is delivered, and finally an intervention phase, for a total of 13 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Trauma Life Support (Experimental): The intervention will be ATLS® training, a proprietary 2.5 day course teaching a standardised approach to trauma patient care using the concepts of a primary and secondary survey. Physicians will be trained in an accredited ATLS® training facility in India.
  Interventions: Behavioral: Advanced Trauma Life Support training
- Standard care (No Intervention): Standard care varies across hospitals in India, but trauma patients are initially managed by casualty medical officers, surgical residents, or emergency medicine residents. They are mainly first- or second-year residents who resuscitate patients, perform interventions and refer patients for imaging or other investigations. Compared with other settings where a trauma team approach is adopted, nurses and other healthcare professionals are only involved to a limited extent during the initial management.

INTERVENTIONS:
Behavioral: Advanced Trauma Life Support training — Advanced Trauma Life Support (ATLS) is a proprietary 2.5 day course teaching a standardised approach to trauma patient care using the concepts of a primary and secondary survey. The programme was developed by the Committee of Trauma of the American College of Surgeons. The course includes intial treatment and resuscitation, triage and interfacility transfers. Leaning is based on practical scenario-driven skill stations, lectures and includes a final performance proficiency evaluation. Physicians will be trained in an accredited ATLS training facility in India.
  Arms: Advanced Trauma Life Support

SUMMARY:
Rationale:

Trauma is a massive global health issue. Many training programmes have been developed to help physicians in the initial management of trauma patients. Among these programmes, Advanced Trauma Life Support® (ATLS®) is the most popular, having trained over one million physicians worldwide. Despite its widespread use, there are no controlled trials showing that ATLS® improves patient outcomes. Multiple systematic reviews emphasise the need for such trials.

Aim:

To compare the effects of ATLS® training with standard care on outcomes in adult trauma patients.

Trial Population:

Adult trauma patients presenting to the emergency department of a participating hospital.

Eligibility Criteria:

Hospitals are secondary or tertiary hospitals in India that admit or refer/transfer for admission at least 400 patients with trauma per year. Clusters are one or more units of physicians providing initial trauma care in the emergency department of tertiary hospitals in India. Patients participants are adult trauma patients who presents to the emergency department of participating hospitals and are admitted or transferred for admission.

Ethical Considerations:

The study will use an opt-out consent approach for in-hospital collection of routinely recorded data, in which consent is presumed unless actively declined. Informed consent for non-routinely recorded data including out of hospital follow up will be obtained. Patients who are unconscious or lack a legally authorized representative will be included under a waiver of informed consent. Note that consent here refers to consent to data collection, as it will not be possible for patients to opt out from being subjected to the intervention. This approach is justified because the trial can be considered to involve only minimal risk and the data collection is non-invasive and mostly involve extracting routinely collected data from medical records.

Funding:

Swedish Research Council (reg. no. 2023-03128), Laerdal Foundation (reg. no. 2023-0297).

Special considerations:

This trial is not yet fully funded. The Trial Management Group has decided to proceed with the trial with the expectation that additional funding will be secured. The Joint Trial Steering and Data Monitoring Committee will be informed of the funding status at each meeting. If funding is not secured, the trial will be stopped. This will likely result in an underpowered trial. The justification for this decision is that the intervention is considered standard of care in many countries and the data collection is considered minimal risk. There is therefore a very small risk of harm to patient participants, but a potential direct benefit to those.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 15 years;
* trauma occurred less than 48 hours before arrival at the hospital;
* present to the emergency department of participating hospitals, with a history of trauma defined as having any of the reasons listed in the International Classification of Diseases chapter XX as the reason for presenting;
* admitted or died between arrival at the hospital and admission, or referred/transferred from the emergency department of a participating hospital to another hospital for admission; and
* managed by a participating cluster in the emergency department.

Exclusion Criteria:

* present with isolated limb injuries; or
* are directly admitted to a ward without being seen by a physician in the emergency department.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4320 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality within 30 days of arrival at the emergency department | 30 days
  Clinical research coordinators will extract information on death from patient hospital records. If the patient has been transferred to another hospital, the clinical research coordinators will collect data on this outcome by calling the patient or a patient representative, or by contacting the hospital to which the patient was transferred. Data on this outcome will be collected continuously during the trial.

CONTACTS AND LOCATIONS:
Locations (10):
- India (10):
  - Assam Medical College & Hospital, Dibrugarh, Assam
  - KEM Hospital, Mumbai, Maharashtra
  - Lokmanya Tilak Municipal General Hospital, Mumbai, Maharashtra
  - Hridaysamrat Balasaheb Thackre Mun. Medical college and Dr. R.N. Cooper Hospital, Mumbai, Maharashtra
  - Holy Family Hospital, New Delhi, New Delhi
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Christian Medical College & Hospital, Ludhiana, Punjab
  - Himalayan Institute of Medical Sciences, Swami Rama Himalayan University, Dehradun, Uttarakhand
  - Institute of Post-Graduate Medical Education and Research and Seth Sukhlal Karnani Memorial Hospital (IPGMER and SSKM Hospital), Kolkata, West Bengal
  - Government Medical College Hospital, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ranjan S, Falth S, Kharat P, Bassi A, Bakhshi GD, Basak D, Berg J, Chatterjee S, Fellander-Tsai L, Hemming K, Jha V, Kasza J, Khajanchi M, Martin J, Mishra A, Olofsson A, Roy N, Singh R, Soni KD, Gerdin Warnberg M. Effects of Advanced Trauma Life Support(R) training compared with standard care on adult trauma patient outcomes (ADVANCE TRAUMA): study protocol for a stepped-wedge cluster randomised trial. Trials. 2026 Feb 3. doi: 10.1186/s13063-026-09491-z. Online ahead of print. PMID 41630085